CLINICAL TRIAL: NCT04968132
Title: Opioid Reduction in Orthopaedic Surgery (OREOS): a Feasibility Randomized Controlled Trial in Knee Replacement Patients
Brief Title: Opioid Reduction in Orthopaedic Surgery (OREOS) - Knees
Acronym: OREOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kim Madden (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); McMaster Surgical Associates (Other); St. Joseph's Healthcare Foundation (Other)
Responsible Party: Sponsor-Investigator, Kim Madden, Assistant Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OREOS-knee
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis; Chronic Post Operative Pain
Keywords: Total knee arthroplasty; education; opioid reduction; cognitive behavioural therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2 group parallel randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study interventions, patients and the health care team cannot be blinded. An independent blinded surgeon will evaluate each adverse event to minimize the risk of bias for that outcome. The primary study outcome of non-opioid pain control will be collected using a daily e-diary up to 8 weeks. Other study outcomes will be collected by a research personnel not involved in the clinical care. Data analysts will be blinded for all outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care group (Active Comparator): This group will receive standard perioperative care, surgical treatment, and pain medications.
  Interventions: Other: Standard care
- Opioid reduction group (Experimental): Patients will participate in a multicomponent pathway coordinated by a trained coordinator who will facilitate patient participation and engagement with each interventional component.
  Interventions: Other: Multicomponent opioid reduction and pain management pathway

INTERVENTIONS:
Other: Multicomponent opioid reduction and pain management pathway — Pre-operative pain education and expectation setting, identification and modification of risk factors in high risk patients, postoperative individualized analgesic prescriptions, and continued support for pan control and recovery facilitated by an interventions coordinator.
  Arms: Opioid reduction group
Other: Standard care — Standard perioperative care, surgical treatment, and pain medications.
  Arms: Standard care group

SUMMARY:
Knee replacements are the second most common surgery in Canada. Most patients recover very well but research consistently shows that 1 in 5 patients still have pain many months after surgery. Doctors often prescribe opioid medications for pain after surgery (e.g. Percocet, hydromorphone, codeine). These medications can be helpful for some people, but they can also be dangerous, particularly when used for a long time. Many patients don't like the way opioids make them feel and would prefer alternative pain management strategies. Some people become addicted to opioids, have a difficult time reducing the dose of opioids, or have lasting health problems after using them.

People in this study will be randomized to either have usual care or a new pathway designed to improve pain control and decrease opioid use after knee replacements. This study will have an intervention coordinator who will assess patients before surgery and who will follow up with patients regularly after surgery to make sure their pain is controlled and to avoid long-term opioid use. This study will use education, physiotherapy, psychological therapy, ice/cold, and non-opioid pain medications. As pain medications may work differently in different patients, the coordinator will check on each patient to look for pain control and assist to reduce the amount of opioids used after surgery.

This study will help people have safer and more effective pain management after surgery which may lead to better recovery, higher satisfaction, and a lower risk of being harmed by opioids after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+)
* Undergoing elective total knee arthroplasty (TKA) for knee arthritis
* Can use a simple electronic (phone or tablet) device
* Provide informed consent to participate

Exclusion Criteria:

* Revision surgery
* Simultaneous bilateral arthroplasties
* Unable to consent (e.g., cognitive disability or substantial language barrier without a support person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Intervention adherence [feasibility] | 8 weeks
  Percentage of patients receiving at least 3 of the 4 trial intervention components.
Participant recruitment [feasibility] | 4 months
  Number of participants recruited
Participant retention [feasibility] | 8 weeks
  Number of participants completing the primary outcome

SECONDARY OUTCOMES:
Opioid-free pain control | 8 weeks
  Three or more consecutive days of <4/10 pain score on a 0-10 numeric rating scale (NRS; lower score is better) with no opioid use for the operated knee.
Chronic post-surgical pain (CPSP) | 12 months
  Defined by the International Classification of Diseases version-11 (ICD-11) criteria
CPSP intensity of resting and movement evoked pain | 12 months
  Measured on a 0-10 numeric rating scale (NRS; lower score is better)
Postoperative opioid use | 12 months
  Presence of daily opioid use, started after surgery or increased after surgery (binary)
Satisfaction with pain control | 12 months
  0 to 100 scale (0=extremely dissatisfied, 100=extremely satisfied)
Health related quality of life | 12 months
  EuroQol-5 Dimensions (EQ-5D)
Complications | 12 months
  Surgery-related and knee-related adverse events, pain medication related adverse events, and readmissions

OTHER OUTCOMES:
Health economics | 12 months
  Investigators will use the EQ-5D to assess health utilities for the purpose of health economic analyses (e.g., cost-effectiveness). Intervention costs and healthcare resource utilization information (e.g., hospitalization, physician visits) as well as information on productivity (e.g., time missed from work) will be collected using a self-administered questionnaire, which will be developed for the purpose of this study

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Shanthanna, MD PhD FRCPC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Madden K, Pallapothu S, Young Shing D, Adili A, Bhandari M, Carlesso L, Khan M, Kleinlugtenbelt YV, Krsmanovic A, Nowakowski M, Packham T, Romeril E, Tarride JE, Thabane L, Tushinski DM, Wallace C, Winemaker M, Shanthanna H. Opioid reduction and enhanced recovery in orthopaedic surgery (OREOS): a protocol for a feasibility randomised controlled trial in patients undergoing total knee arthroplasty. Pilot Feasibility Stud. 2024 Feb 15;10(1):30. doi: 10.1186/s40814-024-01457-9. PMID 38360686